CLINICAL TRIAL: NCT03550014
Title: The Effect of Physical Therapy Interventions Directed at the Low Back Versus Low Back and Hips for Individuals With a Primary Complaint of Low Back Pain: A Randomized Clinical Trial
Brief Title: Effectiveness of Physical Therapy Interventions for Low Back Pain Targeting the Low Back Only or Low Back Plus Hips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of Newcastle, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24664
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain; Hip Disease
Keywords: Low Back Pain; Hip; Physical Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to have receive physical therapy targeting the low back only or low back plus hip(s). Neither the participants or investigators can be blinded during this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Back Only (Active Comparator): Participants randomized to the Low Back Only arm will receive physical therapy as directed by the treating physical therapist targeting the lower back.
  Interventions: Procedure: Low Back Only
- Low Back+Hip (Active Comparator): Participants randomized to the Low Back+Hip arm will receive physical therapy as directed by the treating physical therapist targeting the lower back. In addition to that treatment, participants will received hands-on and exercise physical therapy interventions directed at the hip(s).
  Interventions: Procedure: Low Back+Hip

INTERVENTIONS:
Procedure: Low Back Only — The physical therapy interventions are commonly performed in and may include stretching, strengthening, hands-on techniques, etc. The interventions will only be directed at the lower back. Standard plan of care delivered to participants with low back pain and concurrent hip impairments within scope of licensure.
  Other Names: standard physical therapy care
  Arms: Low Back Only
Procedure: Low Back+Hip — The physical therapy interventions are commonly performed in and may include stretching, strengthening, hands-on techniques, etc. The interventions will be directed at the lower back and the hips. Standard plan of care delivered to participants with low back pain and concurrent hip impairments within scope of licensure.
  Other Names: standard physical therapy care
  Arms: Low Back+Hip

SUMMARY:
Low back pain (LBP) is the leading cause of disability worldwide and has substantial impacts on pain and function for an individual. Some individuals with LBP seek physical therapy for their condition. The purpose of the study is to determine whether individuals with LBP have improved pain and disability following physical therapy targeting either the low back only or low back plus hip(s).

DETAILED DESCRIPTION:
Often, individuals with LBP also have concurrent impairments in strength and/or range of motion of one or both hips. Physical therapists may or may not decide to treat the concurrent hip impairments for an individual with LBP based on their clinical decision making. Currently, it is unknown which approach leads to superior patient outcomes in terms of pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Modified Oswestry Disability Index (ODI) ≥ 20%
* Numeric Pain Rating Scale (NPRS) of ≥ 2 points
* Primary complaint of low back pain with at least one hip impairment in one or both hips

Exclusion Criteria:

* Contraindications to manual therapy
* Severe trauma to the lumbar spine or hip(s) in the last 6 weeks
* 'Red flag' symptoms including:

  * Tumor
  * Metabolic disease
  * Rheumatoid arthritis or other systemic rheumatologic disorders
  * Acute fracture
  * Bowel/Bladder dysfunction
  * Prolonged history of corticosteroid use
  * Evidence of central nervous system involvement
* Two or more positive neurologic signs consistent with nerve root compression:

  * Diminished muscle stretch reflexes of lower extremity
  * Muscle weakness in any lower extremity myotome
  * Diminished or absent sensation in any lower extremity dermatome
* Spinal surgery in the last 6 months
* Total Hip Arthroplasty
* Currently pregnant or post-partum ≤ 6 months
* Osteoporosis
* History of cancer within the last 12 months
* Inability to understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Modified Oswestry Disability Index (ODI) | Baseline, 2 weeks, end of intervention (discharge; an average of 6 weeks), 6 month and 12 months
  The ODI is a reliable and responsive 10 question condition-specific self-report measure for individuals with LBP. The ODI is scored on a scale from 0% to 100%, higher scores indicating higher levels of disability.
Change from baseline on the Numeric Pain Rating Scale (NPRS) | Baseline, 2 weeks, end of intervention (discharge; an average of 6 weeks), 6 month and 12 months
  The NPRS is an 11 point scale (0-10) where the participant is asked to rate their pain intensity at best, worst and average over the last 24 hours. The scale is anchored on the left (score of 0) with the phrase "No Pain" and on the right (score of 10) with the phrase "Worst Imaginable Pain". The NPRS is a valid and reliable assessment of pain severity for individuals with low back pain.

SECONDARY OUTCOMES:
Change from baseline on the Fear Avoidance Beliefs Questionnaire (FABQ) | Baseline, 2 weeks, end of intervention (discharge; an average of 6 weeks), 6 month and 12 months
  The FABQ is a 16-item questionnaire designed to quantify fear and avoidance beliefs in patients with LBP. The FABQ has two sub-scales, a 7-item scale to measure fear-avoidance beliefs about work-related activities (FABQ-W) and a 4-item scale to measure fear-avoidance beliefs about physical activity (FABQ-PA). Each item is scored from 0-6 with possible scores ranging between 0-24 and 0-42 for the physical activity and work subscales, respectively, with higher scores representing increased fear-avoidance beliefs. Recent evidence suggests that the FABQ may be a valuable piece of data for predicting outcomes following intervention in work-related low back pain patients.
Change from baseline on the Global Rating of Change (GROC) | 2 weeks, end of intervention (discharge; an average of 6 weeks), 6 month and 12 months
  The GROC is a 15-point scale that ranges from -7 (a very great deal worse) to zero (about the same) to +7 (a very great deal better). 28 Descriptors of worsening or improving are assigned values from -1 to -6 and +1 to +6 respectively. It has been reported that scores of +4 and +5 are indicative of moderate changes in patient status and scores of +6 and +7 indicate large changes in patient status. This scale will not be administered at baseline evaluation, but at all subsequent time points.
Change from baseline on the Patient Acceptable Symptom State (PASS) | 2 weeks, end of intervention (discharge; an average of 6 weeks), 6 month and 12 months
  The PASS is a single question designed to determine if an individual considers their current status as 'feeling well'. The PASS question was: "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" The participant response with a 'yes' or 'no' answer.
Change from baseline on the Godin Leisure-Time Physical Activity Questionnaire | Baseline, end of intervention (discharge; an average of 6 weeks)
  The Godin-Shepard Leisure-Time Physical Activity Questionnaire allows for self-reported leisure-time physical activity. It allows the participant to designate the number of times per week that the engage in physical activities that are of varying intensities (strenuous, moderate, mild). The sum of each intensity is then multiplied by their corresponding metabolic equivalent values of 9, 5, and 3, respectively. High total scores provide the frequency and intensity of exercise that an individual participates in on a weekly basis. The questionnaire has been validated for classifying healthy adults into active and insufficiently active categories. A lack of physical activity in leisure times have been associated with increased prevalence of low back pain.
Patient Health Questionnaire-2 (PHQ-2) | Baseline
  The PHQ-2 is a validated two-question screening questionnaire that is used to determine the presence of depressive disorders. Individuals with low back pain that have depressive symptoms tend to have poor outcomes. The two questions are completed by the participant and scored on a 0-3 scale. The scores for both questions are summed with a cut off score of 3 or higher is considered more at risk for the presence of any depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Burns, DPT, Principal Investigator — Temple University; Suzanne J Snodgrass, PhD, Study Chair — The University of Newcastle; Darren A Rivett, PhD, Study Director — The University of Newcastle; Joshua A Cleland, DPT, PhD, Study Director — Franklin Pierce University
Locations (7):
- United States (7):
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Franciscan Health Sports Medicine Physical Therapy Clinic, Indianapolis, Indiana
  - BSR Physical Therapy, Barnegat, New Jersey
  - BSR Physical Therapy, Manahawkin, New Jersey
  - Kinetic Physical Therapy, Collegeville, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Bellin Health Systems, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No
All data will be used as part of research project for dissertation purposes and not shared to other researchers

REFERENCES:
- [Derived] Burns SA, Cleland JA, Rivett DA, Snodgrass SJ. Effectiveness of physical therapy interventions for low back pain targeting the low back only or low back plus hips: a randomized controlled trial protocol. Braz J Phys Ther. 2018 Sep-Oct;22(5):424-430. doi: 10.1016/j.bjpt.2018.08.014. Epub 2018 Sep 7. PMID 30217693